CLINICAL TRIAL: NCT04321499
Title: Establishing a Non-invasive Diagnostic Biomarker Test for Early Diagnosis of Lung Cancer
Brief Title: SHOX2_PTGER4 DNA Methlyation in Lung Cancer
Acronym: Epi1
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Kaid Darwiche, Priv.-Doz. Dr. med. Kaid Darwiche, head of department of interventional pneumology, University Hospital, Essen
Other Study IDs: SHOX2 and PTGER4
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Lungcancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- lung cancer: stage IA-IIIA lung cancer
  Interventions: Genetic: lung cancer
- benign nodules: ruled out lung cancer via Operation or CT-scan follow-up
  Interventions: Genetic: lung cancer

INTERVENTIONS:
Genetic: lung cancer — PCR for SHOX2 and PTGER4

SUMMARY:
Data on SHOX2 and PTGER4 DNA Methylation suggest possible use as a biomarker for early lung cancer diagnosis.

In this study a control group consisting of COPD patients with a CT-scan of the chest no older than 6 weeks and a control group of patients with a nodule and ruled out diagnosis of lung cancer will be included.

SHOX2 and PTGER4 will be analyzed via PCR.

DETAILED DESCRIPTION:
Data on SHOX2 and PTGER4 DNA Methylation suggest possible use as a biomarker for early lung cancer diagnosis.

In this study a control group consisting of COPD patients with a CT-scan of the chest no older than 6 weeks and a control group of patients with a nodule and ruled out diagnosis of lung cancer will be included.

A total of 150 patients will be enrolled in this study. SHOX2 and PTGER4 will be analyzed via PCR of blood plasma samples.

ELIGIBILITY:
Inclusion Criteria:

suspicious finding for lung cancer on CT-scan

Exclusion Criteria:

* history significant for former malignant diseases

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung cancer, benign nodule
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
DNA Methylation at early stages of lung cancer | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kaid Darwiche, MD, Principal Investigator — head of deparment of interventional pneumology, Ruhrlandklinik, UHEssen
Locations (1):
- Ruhrlandklinik, Department of Interventional Pneumology, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiss G, Schlegel A, Kottwitz D, Konig T, Tetzner R. Validation of the SHOX2/PTGER4 DNA Methylation Marker Panel for Plasma-Based Discrimination between Patients with Malignant and Nonmalignant Lung Disease. J Thorac Oncol. 2017 Jan;12(1):77-84. doi: 10.1016/j.jtho.2016.08.123. Epub 2016 Aug 18. PMID 27544059